CLINICAL TRIAL: NCT04392232
Title: A Phase 2 Study of COVID 19 Convalescent Plasma in High Risk Patients With COVID 19 Infection
Brief Title: A Study of COVID 19 Convalescent Plasma in High Risk Patients With COVID 19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-045
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus; COVID-19; Convalescent Plasma
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Non-Randomized, single arm study of convalescent plasma treatment of covid 19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Convalescent Plasma (Experimental)
  Interventions: Drug: Convalescent Plasma

INTERVENTIONS:
Drug: Convalescent Plasma — • Investigational Product
  o COVID-19 convalescent plasma will be obtained from an FDA-registered blood establishment (Hoxworth) that follows donor eligibility criteria and donor qualifications as outlined in section III.C.I of the Investigational COVID-19 Convalescent Plasma Guidance for Industry.

SUMMARY:
Purpose of Study

• The purpose of this study to evaluate, the effectiveness of convalescent plasma in combatting the symptoms and effects of the coronavirus disease, COVID-19. Beyond supportive care, there are no proven treatment options for COVID-19.

DETAILED DESCRIPTION:
Hypothesis or Research Question • Is convalescent plasma from patients previously infected with COVID-19 an effective treatment option for high risk patients through the utilization of passive immunity?

o Is the mortality rate reduced through the use of this treatment?

Background Passive antibody therapy involves the administration of antibodies to a given agent to a susceptible individual for the purpose of preventing or treating an infectious disease due to that agent. In contrast, active vaccination requires the induction of an immune response that takes time to develop and varies depending on the vaccine recipient. Some immunocompromised patients fail to achieve an adequate immune response. Thus, passive antibody administration is the only means of providing immediate immunity to susceptible persons and immunity of any measurable kind for highly immunocompromised patients.

Passive antibody therapy has a storied history going back to the 1890s and was the only means of treating certain infectious diseases prior to the development of antimicrobial therapy in the 1940s (1,2). Experience from prior outbreaks with other coronaviruses, such as SARS-CoV-1 shows that such convalescent plasma contains neutralizing antibodies to the relevant virus (3). In the case of SARS-CoV-2, the anticipated mechanism of action by which passive antibody therapy would mediate protection is viral neutralization. However, other mechanisms may be possible, such as antibody dependent cellular cytotoxicity and/or phagocytosis. Convalescent serum was also used in the 2013 African Ebola epidemic. A small non-randomized study in Sierra Leone revealed a significant increase in survival for those treated with convalescent whole blood relative to those who received standard treatment (4).

The only antibody type that is currently available for immediate use is that found in human convalescent plasma. As more individuals contract COVID-19 and recover, the number of potential donors will continue to increase.

A general principle of passive antibody therapy is that it is more effective when used for prophylaxis than for treatment of disease. When used for therapy, antibody is most effective when administered shortly after the onset of symptoms. The reason for temporal variation in efficacy is not well understood but could reflect that passive antibody works by neutralizing the initial inoculum, which is likely to be much smaller than that of established disease. Another explanation is that antibody works by modifying the inflammatory response, which is also easier during the initial immune response, which may be asymptomatic (5). As an example, passive antibody therapy for pneumococcal pneumonia was most effective when administered shortly after the onset of symptoms and there was no benefit if antibody administration was delayed past the third day of disease (6). In this context, we seek to treat patients who are sick enough to warrant hospitalization but prior to the onset of overwhelming disease including advanced systemic inflammatory response, sepsis, and/or ARDS. We hypothesize that convalescent plasma will be more effective given earlier in the hospital course and we aim to maximize the overall potential population benefit by directing the plasma to patients who at presentation are predicted to be at high risk but before they are in advanced overwhelming disease. We aim to start plasma therapy within 24 hours of admission or when high risk features are first evident.

For passive antibody therapy to be effective, a sufficient amount of antibody must be administered. When given to a susceptible person, this antibody will circulate in the blood, reach tissues and provide protection against infection. Depending on the antibody amount and composition, the protection conferred by the transferred immunoglobulin can last from weeks to months.

In the 21st century, there were two other epidemics with coronaviruses that were associated with high mortality, SARS1 in 2003 and MERS in 2012. In both outbreaks, the high mortality and absence of effective therapies led to the use of convalescent plasma. The largest study involved the treatment of 80 patients in Hong Kong with SARS (7). Patients treated before day 14 had improved prognosis defined by discharge from hospital before day 22, consistent with the notion that earlier administration is more likely to be effective. In addition, those who were RT-PCR positive and seronegative for coronavirus at the time of therapy had improved prognosis. There is also some anecdotal information on the use of convalescent plasma in seriously ill individuals. Three patients with SARS in Taiwan were treated with 500 ml of convalescent plasma, resulting in a reduction in plasma virus titer and each survived (8). Three patients with MERS in South Korea were treated with convalescent plasma, but only two of the recipients had neutralizing antibody in their plasma (9). The latter study highlights a challenge in using convalescent plasma, namely, that some who recover from viral disease may not have high titers of neutralizing antibody (10). Consistent with this point, an analysis of 99 samples of convalescent sera from patients with MERS showed that 87 had neutralizing antibody with a geometric mean titer of 1:61. This suggests that antibody declines with time and/or that few patients make high titer responses.

It is also possible that other types of non-neutralizing antibodies are made that contribute to protection and recovery as described for other viral diseases (11). There are reports that convalescent plasma was used for therapy of patients with COVID-19 in China during the current outbreak (http://www.xinhuanet.com/english/2020-02/28/c_138828177.htm). Although few details are available from the Chinese experience and published studies involved small numbers of patients, the available information suggests that convalescent plasma administration reduces viral load and was safe.

ELIGIBILITY:
• Eligibility Criteria

* Participants will be 16 years or older.
* COVID-19 infection demonstrated via SARS-CoV-2 PCR testing.
* Admitted to the hospital for treatment of Covid 19.
* Patients must have severe/high risk disease as defined by the presence of any one of the following:

Respiratory frequency ≥ 25/minute Oxygen saturation ≤ 93% on room air Partial pressure of arterial oxygen to fraction of inspired oxygen ration < 300, or pulse oximetric saturation to fraction of inspired oxygen ratio < 315.

Lung infiltrates > 50% within 24-48 hours of admission on Chest X-Ray or, Ferritin > 1000 or absolute lymphocyte count < 600 or D-Dimer > 1.00

* ABO Blood Type available.
* Pregnant women will be permitted to participate in this study.

  • Exclusion criteria
* Previous history of life threatening or severe adverse reactions to transfusion blood products..

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Survival Rate | At 28 Days
  % patients who survived

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Coyle, MD, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No